CLINICAL TRIAL: NCT01701570
Title: Mediators of Perceived Exercise Effort in Type 2 Diabetes - Barriers to Physical Activity
Brief Title: Barriers to Physical Activity in People With Type 2 Diabetes
Acronym: Rxercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0909; 6147 (Other: University of Colorado CTRC)
Record Dates: First submitted 2012-06-13; First posted 2012-10-05 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Exercise; Rate of Perceived Exertion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- An Active Comparator exercise training intervention (Active Comparator): The Active Comparator Groupwill participate in an exercise training intervention to distinguish the relative roles of objective factors (lactate level) and subjective factors (self-efficacy) in mediating pre-post change in RPE during low, moderate, and vigorous exercise.
  Interventions: Other: Supervised Exercise Training
- A Placebo Attention Control (Placebo Comparator): The placebo attention control group will receive monthly diabetes education and phone calls phone calls to monitor their blood glucose levels. Participants will receive an accelerometer to wear for one week.
  Interventions: Behavioral: Placebo Attention Control

INTERVENTIONS:
Behavioral: Placebo Attention Control — The placebo attention control group will receive weekly phone calls to monitor their blood glucose levels.
  Arms: A Placebo Attention Control
Other: Supervised Exercise Training — The 20-week aerobic exercise training intervention provides supervised exercise training sessions 3 times weekly following the HERITAGE study training model that was feasible in prior studies with older, sedentary overweight adults (55%maximal oxygen uptake (VO2max) for 30 minutes per session at study entry with progressive titration to 70-80% VO2max for 50 minutes).
  Arms: An Active Comparator exercise training intervention

SUMMARY:
The investigators plan to learn more about how different levels of exercise feel to people with Type 2 Diabetes and how it feels to people without Type 2 Diabetes. This study team will also look at what causes exercise to feel harder or easier to people with and without Type 2 Diabetes. The investigators will also compare the potential benefits of supervised exercise training to that of diabetes education/blood sugar monitoring.

DETAILED DESCRIPTION:
Exercise is a potent therapy to reduce cardiovascular mortality in Type 2 Diabetes (T2D). Although exercise is a cornerstone of treatment for T2D, people with T2D are more sedentary than similarly obese people without diabetes, for reasons that are unclear. Interventions which combined behavioral support and physical activity prescriptions successfully increased physical activity levels for people with T2D and at-risk for T2D. However, the program components which mediated increased physical activity were combined and thus the individual benefits of each component remain unknown. Given the success of these combined programs, it appears behavioral support and other psychological factors may play an important role. The study investigators are interested in the predictors of physical activity adherence in T2D as key targets for future interventions.

One likely factor which may influence physical activity adherence is perceived exercise effort. The study investigators reported, based on a small study, that perceived exercise effort is worse in people with T2D than in healthy obese controls, as measured by the Borg Rating of Perceived Exertion (RPE), even during low intensity exercise. Thus, one strategy to increase physical activity in T2D is to first identify the mediators of RPE in the proposed study and then to address them in future studies. The preliminary data suggest that likely mediators of RPE are both objective and subjective in nature. A key objective mediator of RPE is serum lactate level during exercise, which is a physiological marker of effort, and is disproportionately elevated in people with T2D vs. healthy controls. A key subjective mediator of RPE is self-efficacy, which influences the perception of exercise effort, and is disproportionately worse in people with T2D vs. healthy controls. To develop optimal physical activity interventions for people with T2D, the study investigators must understand whether RPE differences vary across the spectrum of exercise intensities (Aim 1), and the investigators must also determine the mediators of RPE across exercise intensities (Aim 2). Mediators of RPE in low-to-moderate intensity exercise are particularly important, because walking is a preferred physical activity for people with T2D.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary men and women not participating in a regular exercise program (> 60 minutes of exercise per week)
* If subject has diabetes,

  * must be uncomplicated type 2 diabetes (T2D) and
  * <15 years since T2D diagnosis.
* Ages of 50-70 years
* BMI between 25 and 35
* Subjects can only be taking the following oral hypoglycemic drugs:

  * metformin,
  * sulfonylureas or
  * sitagliptin.
* Persons with T2D only if they have total glycosylated hemoglobin levels (HbA1C) <8.0% (adequate control) on therapy.
* Control subjects must have:

  * HbA1C < 5.7% and
  * a fasting blood glucose of <100 mg/dl suggesting no significant insulin resistance.
* All women must be post-menopausal, documented by menstrual history and follicle stimulating hormone (FSH) level.
* Those who have quit smoking for at least 1 year will be accepted.
* Absence of comorbid conditions that could affect exercise will be confirmed by history, physical examination and laboratory testing.

Exclusion Criteria:

* Persons with clinically evident distal symmetrical neuropathy, determined by evaluation of symptoms (numbness, paresthesia) and signs (elicited by vibration, pinprick, light touch, ankle jerks), will be excluded from further study as neuropathy may limit exercise performance.

  * Specifically, if monofilament sensation is absent at the level of the ankles, then participants will be excluded from study participation.
* Persons with autonomic dysfunction (>20 mm fall in upright BP without a change in heart rate) will be excluded as well, due to associated limitations of exercise performance.
* Current use of insulin or other oral hypoglycemic medications.
* Current smokers will be excluded since smoking can impair cardiovascular (CV) exercise performance
* Persons will be excluded if they have:

  * evidence of heart disease by history (Prior heart attack or bypass surgery, heart failure, or significant valvular disease) or
  * abnormal resting electrocardiogram (EKG) consistent with prior infarct or latent ischemia (unless cardiovascular stress imaging or catheterization shows they do not have coronary artery disease).
  * left or right bundle branch block on resting EKG (precludes recognition of ischemic EKG changes with exercise) or
  * abnormal exercise EKG (> 1 mm ST segment depression 80 msec out in the ST segment for 3 consecutive beats).
* Persons with angina or any other exercise-limiting cardiovascular, pulmonary or musculoskeletal symptoms.
* Presence of:

  * systolic blood pressure >145 mm Hg at rest or >250 mm Hg with exercise or
  * diastolic blood pressure >90 mm Hg at rest or >115 mm Hg with exercise.
* Subjects with:

  * proteinuria (urine protein >220 mg/dl) or
  * creatinine > 1.6 mg/dl, suggestive of renal disease.
* Subjects with:

  * total cholesterol >220 mg/dl,
  * low density lipoprotein > 130 mg/dl, or
  * triglycerides > 250 mg/dl, will be excluded given the potential insulin resistance and endothelial dysfunction associated with these cholesterol parameters.
* Control subjects who have more than two immediate family members with type 2 diabetes.
* Chronic obstructive pulmonary disease demonstrated by a ratio of

  * Forced Expiratory Volume in 1 second (FEV1),
  * Forced Vital Capacity (FVC) < 0.70, or
  * FEV1 <70% predicted during spirometry.
* Persons weighing more than 300 pounds will be excluded as this exceeds the weight capacity of our Dual Energy X-ray Absorptiometry device
* Participants with moderate cognitive impairment (Folstein Mini-Mental Status Examination (MMSE) score <24).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Rating of perceived exercise effort (RPE) during exercise (Borg RPE scale) | Baseline, week 20
  RPE was developed by Dr. Gunnar Borg and is a validated, self-reported measure of perceived effort during exercise. Possible scores range from 6 (no effort, resting) to 20 (maximal effort). Change = RPE post-intervention (week 20) - RPE baseline.

SECONDARY OUTCOMES:
Serum lactate during exercise | Baseline, week 20
  Serum lactate is measured by the University of Colorado clinical laboratory (Units = mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Huebschmann, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States